CLINICAL TRIAL: NCT07366320
Title: Effects of Four-Week Rhodiola Rosea Supplementation on Physical Fitness, Neuromuscular Performance and Decision-Making in Competitive Football Players: A Randomised Controlled Trial
Brief Title: Effects of Four-Week Rhodiola Rosea Supplementation on Physical Fitness, Neuromuscular Performance, and Decision-Making in Competitive Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Principal Investigator, Yue Dou, Graduate Student, Beijing Sport University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025619H
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Physical Performance and Fatigue in Competitive Football Players
Keywords: Rhodiola rosea; Soccer; Football players; Dietary supplement; Repeated sprint ability; Decision making; Fatigue; Randomized controlled trial
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either Rhodiola rosea supplementation or placebo in a parallel two-arm design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and outcome assessors were blinded to group allocation. Supplements and placebo were identical in appearance and packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhodiola rosea Group (Experimental): Participants received Rhodiola rosea supplementation for 4 weeks in addition to their regular football training.
  Interventions: Dietary Supplement: Rhodiola rosea extract
- Placebo (Placebo Comparator): Participants consumed placebo capsules identical in appearance to Rhodiola rosea for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Rhodiola rosea extract — Participants assigned to this intervention will receive Rhodiola rosea extract for 4 weeks in addition to their regular football training. The supplement will be administered orally in capsule form at a dose of 2,400 mg per day, given twice daily. The extract is standardized to salidroside, providing a total of 12 mg salidroside per daily dose. The capsules contain starch as excipient and gelatin as the capsule shell. All supplements are sourced from the same production batch to ensure consistency throughout the intervention period. Adherence will be monitored by capsule count and compliance logs.
  Other Names: Rhodiola
  Arms: Rhodiola rosea Group
Other: Placebo — Participants assigned to this intervention will receive placebo capsules identical in appearance, taste, and packaging to the Rhodiola rosea capsules for 4 weeks in addition to their regular football training. The placebo contains inert ingredients and is administered orally following the same dosing schedule as the Rhodiola rosea group.
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
This study investigates whether four weeks of Rhodiola rosea supplementation can improve physical fitness, neuromuscular performance, and decision-making ability in competitive male football players. Participants are randomly assigned to receive either Rhodiola rosea or a placebo while continuing their regular football training. Before and after the four-week intervention, all participants complete a series of tests, including aerobic fitness, repeated sprint ability, jumping performance, reaction time, and soccer-specific decision-making tasks. Blood samples are also collected to assess fatigue and recovery-related markers. The purpose of this study is to determine whether Rhodiola rosea supplementation can enhance performance and cognitive function under high-intensity training and competition conditions.

DETAILED DESCRIPTION:
This study is a prospective, double-blind supplementation study conducted in competitive male football players to examine the effects of short-term Rhodiola rosea intake on physical and cognitive performance under regular training conditions.

Participants continue their habitual football training while receiving either Rhodiola rosea supplementation or a placebo for four weeks. Performance assessments are conducted before and after the intervention period under standardized conditions.

The study aims to explore whether Rhodiola rosea supplementation may support adaptations related to high-intensity exercise performance, neuromuscular function, and decision-making ability in competitive football players.

ELIGIBILITY:
Inclusion Criteria:

* Male competitive football players aged 18-30 years
* Regular participation in structured football training (≥3 sessions per week)
* Free from musculoskeletal injury for at least 3 months prior to the study
* Not using any nutritional supplements or ergogenic aids for at least 4 weeks before enrollment
* Willing to maintain habitual diet and training throughout the study
* Provided written informed consent

Exclusion Criteria:

* History of cardiovascular, metabolic, neurological, or endocrine disease
* Use of Rhodiola rosea, caffeine, or other performance-enhancing supplements within the past 4 weeks
* Current smoking or substance abuse
* Known allergy to herbal supplements
* Any injury or illness that could affect physical performance or safe participation

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Yo-Yo Intermittent Recovery Test Level 2 (Yo-Yo IR2) distance | Time Frame: Baseline and Week 4
  The Yo-Yo Intermittent Recovery Test Level 2 (Yo-Yo IR2) will be used to assess high-intensity intermittent endurance capacity. The total distance completed during the test will be recorded at baseline and after 4 weeks of Rhodiola rosea or placebo supplementation.

SECONDARY OUTCOMES:
Best sprint time during repeated sprint test | Time Frame: Baseline and Week 4
  Best sprint time (seconds) recorded during a 6 × 30 m repeated sprint test.
Mean sprint time during repeated sprint test | Baseline and Week 4
  Mean sprint time (seconds) calculated across all sprints during a 6 × 30 m repeated sprint test.
Countermovement jump (CMJ) height | Time Frame: Baseline and Week 4
  Vertical jump height will be measured using a countermovement jump test to evaluate lower-limb neuromuscular performance before and after the intervention.
Decision-making reaction time | Time Frame: Baseline and Week 4
  Reaction time (milliseconds) measured during a computer-based soccer-specific decision-making task. Lower values indicate faster responses.
Blood lactate concentration immediately post-repeated sprint exercise | Baseline and Week 4 (immediately post-repeated sprint exercise)
  Capillary blood lactate concentration (mmol/L) measured immediately following a repeated sprint exercise to assess acute metabolic stress.
Decision-making response accuracy | Baseline and Week 4
  Response accuracy (%) measured during a computer-based soccer-specific decision-making task. Higher values indicate better performance.
Blood lactate concentration 3 minutes post-repeated sprint exercise | Baseline and Week 4 (3 minutes post-repeated sprint exercise)
  Capillary blood lactate concentration (mmol/L) measured 3 minutes following a repeated sprint exercise to assess early recovery.
Blood lactate concentration 5 minutes post-repeated sprint exercise | Baseline and Week 4 (5 minutes post-repeated sprint exercise)
  Capillary blood lactate concentration (mmol/L) measured 5 minutes following a repeated sprint exercise to assess late recovery.
Hemoglobin concentration | Time Frame: Baseline and Week 4
  Resting hemoglobin concentration (g/L) measured to assess oxygen-carrying capacity.
Hematocrit | Baseline and Week 4
  Resting hematocrit (%) measured to assess oxygen-carrying capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Dingmeng Ren, PhD, Principal Investigator — Beijing Sport University
Locations (1):
- China Football Institute, Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant confidentiality and institutional data protection policies.